CLINICAL TRIAL: NCT06088134
Title: Urology Department of the First Affiliated Hospital of Chongqing Medical University
Brief Title: Contrast-enhanced CT-based Deep Learning Model for Preoperative Prediction of Disease-free Survival (DFS) in Localized Clear Cell Renal Cell Carcinoma (ccRCC)
Status: Recruiting | Type: Observational
Sponsor: Mingzhao Xiao (Other)
Responsible Party: Sponsor-Investigator, Mingzhao Xiao, Urology Department, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: DL-ccRCC
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Clear Cell Renal Cell Carcinoma; Prognostic Cancer Model; Recurrent Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Non-recurrence group
- Recurrence group

SUMMARY:
This study aims to preoperatively predict DFS of patients with localised ccRCC using a deep learning prognostic model based on enhanced contrast CT images, validate it's predictive ability in multicentre data and compare it's predictive ability with traditional models.

ELIGIBILITY:
Inclusion Criteria:

* underwent partial/radical nephrectomies
* histologically diagnosed as ccRCC
* with complete clinical data and preoperative CT image data

Exclusion Criteria:

* with incomplete clinic-pathological data
* lack of preoperative contrast-enhanced CT images or the image quality was unsuitable for analysis
* who received pre-surgery neoadjuvant or adjuvant therapies
* with multiple renal tumors or/and had synchronous metastasis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted to urology departments at participating medical centres
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | recruitment occurred between June 2013 and March 2020
  the interval from the date of surgery to disease recurrence, all-cause mortality or the last visit

CONTACTS AND LOCATIONS:
Locations (1):
- Yingjie Xv, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xv Y, Wei Z, Jiang Q, Zhang X, Chen Y, Xiao B, Yin S, Xia Z, Qiu M, Li Y, Tan H, Xiao M. Three-dimensional deep learning model complements existing models for preoperative disease-free survival prediction in localized clear cell renal cell carcinoma: a multicenter retrospective cohort study. Int J Surg. 2024 Nov 1;110(11):7034-7046. doi: 10.1097/JS9.0000000000001808. PMID 38896853